CLINICAL TRIAL: NCT03462342
Title: Combination ATR and PARP Inhibitor (CAPRI) Trial With AZD 6738 and Olaparib in Recurrent Ovarian Cancer
Brief Title: Combination ATR and PARP Inhibitor (CAPRI) Trial With AZD6738 and Olaparib in Recurrent Ovarian Cancer
Acronym: CAPRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 827744, ESR-16-12311
Record Dates: First submitted 2018-02-09; First posted 2018-03-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: High Grade Serous Carcinoma
MeSH Terms: interventions — olaparib; ceralasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- A. Olaparib Pill + AZD6738. (Experimental): Cohort A: Recurrent platinum-sensitive ovarian cancer (progression greater than 6 months from last receipt of platinum-based chemotherapy), approximately 37 patients could be treated with an interim analysis after 17 subjects.
  All patients will receive the combination of AZD6738 and olaparib. Patients will be administered olaparib orally twice daily at 300 mg BD. Patients will be administered AZD6738 orally once daily at 160 mg on days 1 to 7.
  For ease of administration, the AZD6738 should be administered at the same time as one of the olaparib doses and thus with one glass of water.
  Interventions: Drug: Olaparib Pill; Drug: AZD6738
- B. Olaparib Pill + AZD6738. (Experimental): Cohort B: Recurrent platinum-resistant ovarian cancer (progression less than or equal to 6 months of the last receipt), approximately 37 patients could be treated with an interim analysis after 12 subjects.
  All patients will receive the combination of AZD6738 and olaparib. Patients will be administered olaparib orally twice daily at 300 mg BD. Patients will be administered AZD6738 orally once daily at 160 mg on days 1 to 7.
  For ease of administration, the AZD6738 should be administered at the same time as one of the olaparib doses and thus with one glass of water.
  Interventions: Drug: Olaparib Pill; Drug: AZD6738
- C. Olaparib Pill + AZD6738. (Experimental): Cohort C: PARP inhibitor (PARPi) resistant (subjects who have progressed on a PARPi), patients must be platinum-sensitive, and have a germline or somatic BRCA mutation or an HRD mutation. Approximately 12 subjects could be treated.
  All patients will receive the combination of AZD6738 and olaparib. Patients will be administered olaparib orally twice daily at 300 mg BD. Patients will be administered AZD6738 orally once daily at 160 mg on days 1 to 7.
  For ease of administration, the AZD6738 should be administered at the same time as one of the olaparib doses and thus with one glass of water.
  Interventions: Drug: Olaparib Pill; Drug: AZD6738
- D-1. Olaparib Pill + AZD6738. (Experimental): Cohort D Part I: Patients will be platinum sensitive/platinum resistant ovarian cancer. Patient may or may not have received prior PARPi and will be enrolled irrespective of their BRCA status. The number of subjects treated will depend on the number of dose levels explored with a minimum of 12 subjects up to 30 subjects.
  All patients will receive the combination of AZD6738 and olaparib. Cohort D will take a lower dose of olaparib (100-200 mg daily for a 28-day cycle) and a higher dose of AZD6738 (160-320 mg daily for about 14 days). Three to five dosing schedules will be evaluated.
  Interventions: Drug: Olaparib Pill; Drug: AZD6738
- D-2 Olaparib Pill + AZD6738. (Experimental): Cohort D Part II: Patients with ovarian cancer who are PARP inhibitor (PARPi) resistant (patients who have progressed on a PARPi). Patients must be platinum-sensitive and have a germline or somatic BRCA mutation or an HRD mutation. Approximately 12 patients will be treated.
  All patients will receive the combination of AZD6738 and olaparib. Cohort D will take a lower dose of olaparib (100-200 mg daily for a 28-day cycle) and a higher dose of AZD6738 (160-320 mg daily for about 14 days). Three to five dosing schedules will be evaluated.
  Interventions: Drug: Olaparib Pill; Drug: AZD6738

INTERVENTIONS:
Drug: Olaparib Pill — For Cohorts A, B, and C: 300 mg twice daily by mouth which is taken continuously for 28 days, which is one cycle.
  Cohort D 1-2: prescribed lower dose of olaparib (100-200mg daily for a 28-day cycle). Three to five dosing schedules will be evaluated. Dose Levels 1-3: olaparib 100 mg twice daily, Days 1-28. For Dose Levels 4-5: 100-200 mg twice daily, Days 1-28. Other dose levels may be considered and will not exceed AZD6738 160mg twice daily by mouth and olaparib 150mg twice daily by mouth.
  Other Names: Lynparza
Drug: AZD6738 — For Cohorts A, B, and C: 160 mg orally once daily for first 7 days of every cycle (Days 1-7 of each 28-day cycle).
  Cohort D 1-2: Prescribed higher dose of AZD6738 (120-320 mg daily for about 14 days). Three to five dosing schedules will be evaluated.
  Dose Levels 1-3: 120-160 mg twice daily, Days 1-14, in combination with olaparib twice daily, Days 1-28. Alternatively, AZD6738 at 160 mg once daily Days 1-14 with olaparib at 100-150 mg Days 1-28 may be evaluated.
  Dose Levels 4-5: Alternative dosing schedule of AZD6738 at 80-160 mg once or twice daily, weekly intermittent schedule (Days 1-5, 8-12, 15-19) in combination with olaparib 100-200 mg twice daily, Days 1-28 may be evaluated. AZD6738 at 160 mg twice daily, Days 1-7 or 240 mg once daily Days 1-14 with olaparib 100-200 mg twice daily Days 1-28 may be evaluated.
  Other dose levels may be considered and will not exceed AZD6738 160mg twice daily by mouth and olaparib 150mg twice daily by mouth.

SUMMARY:
Investigational agent, AZD6738 will be given in combination with Olaparib to women with recurrent ovarian cancer (platinum-sensitive or platinum-resistant).

This study will determine if using Olaparib in combination with AZD6738 is safe and tolerable and also determine the objective response rate and progression free survival of combination of AZD6738 and Olaparib in women with recurrent ovarian cancer in distinct platinum-sensitive and platinum-resistant cohorts.

ELIGIBILITY:
Inclusion criteria:

For inclusion in the study, patients must fulfill the following criteria:

1. Patients ≥ 18 years of age
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and a life expectancy of at least 6 months.
3. For Cohorts A-C, and Cohort D, Part II, patients must have high grade serous ovarian, primary peritoneal, and/or fallopian tube cancer histologically or cytologically confirmed that is recurrent and for which standard curative measures do not exist or are no longer effective. For Cohort D, Part I, patients may have any non-mucinous epithelial ovarian cancer (including histologies such as clear cell, or endometrioid). Pathology must be reviewed internally at the University of Pennsylvania, Johns Hopkins University, or Harvard University prior to initiation of treatment.
4. All patients under consideration for Cohorts A, B, C, and D, must be willing to undergo mandatory tumor biopsies (non-target lesion). Patients should have at least one lesion (non-target) for biopsy. However, for patients in Cohorts A, B, C, and D, if patients are found to not have a safe lesion to biopsy by the radiology team, they may still be enrolled in the study and forego the biopsy. Patients who undergo attempted biopsies that are unsuccessful may still enroll and receive study drug.
5. All patients must have a measurable disease by RECIST v1.1.
6. Germline BRCA mutation status:

   * Cohorts A and B: Patients with unknown BRCA status or negative BRCA germline mutation status will be permitted to enroll in the study. Patients with known BRCA germline mutations will be permitted to enroll up to a maximum of 10 subjects per cohort.
   * Cohort C and Cohort D Part II: All subjects must have either a germline or somatic BRCA mutation, or other HRD mutation, or tumor is HRD positive. Other HRD mutations will be reviewed for consideration for enrollment by study review committee or University of Pennsylvania principal investigator.
   * Cohort D Part I: Patients will be enrolled irrespective of BRCA status.
7. Adequate renal function, defined as measured creatinine clearance ≥ 51 ml/min.
8. Adequate hepatic function, defined as AST and ALT levels ≤ 2.5 X ULN (for subjects with liver metastases, AST or ALT ≤ 5 × ULN) and total bilirubin < 1.5 X ULN, absent Gilbert's disease.
9. Adequate bone marrow function, defined as absolute neutrophil count (ANC ≥ 1.5 X 109/L), platelet count ≥ 100 x 109/L, and hemoglobin ≥ 10 g/dL (in the absence of transfusion within 28 days prior to dosing).
10. Patients must be at least 2 weeks from previous therapy for their ovarian cancer (chemotherapy, hormonal therapy, and radiation therapy, or investigational agents; 6 weeks for mitomycin C) to initiate screening and 3 weeks from previous therapy to initiate treatment. Hormones for breast cancer management may be continued at the discretion of the provider.
11. Platinum-sensitive is defined as recurrence >6 months by RECIST 1.1 imaging from last platinum. Platinum-resistant is defined as recurrence ≤ 6 months by RECIST 1.1 imaging from last platinum regimen).

    * For Cohort A, there is no limit to number of prior regimens.
    * For Cohort B, patients may not have had more than 3 prior cytotoxic therapies since the development of platinum-resistance.
    * Patients for Cohort D, Part I (dose escalation), patients may be either platinum-sensitive with no limit on prior regimens. Platinum-resistant patients are eligible but they may not have received more than 3 prior cytotoxic therapies since development of platinum resistance.
    * Cohort C and Cohort D, Part II, patients must be platinum-sensitive BUT with no limit to number of prior cytotoxic therapies. These patients must demonstrate adequate bone marrow function as determined by the treating physician.
12. Prior treatment with a PARPi is permitted but not mandatory for Cohorts A and B and Cohort D Part I. Prior treatment with PARPi is mandatory for Cohort C and D Part II. If a patient has received a prior PARPi, then the patient must have demonstrated a clinical benefit of PARPi treatment by an initial response (by CA-125 or imaging) to PARPi treatment or clinical benefit from PARPi treatment as maintenance therapy followed by disease progression for enrollment onto Cohort C and D Part II. Clinical benefit for maintenance is defined as:

    1. prior maintenance with PARPi after 1st line chemotherapy of at least 12 months or
    2. prior maintenance with PARPi after >1 line of chemotherapy for minimum of 6 months. Subjects on Cohort A may have received treatment with PARPi, clinically benefitted, but not have progressed on a PARPi. This arm is to evaluate participants who have received prior PARPi (PARPi after PARPi).

    If the prior PARP inhibitor used was olaparib, it must have been tolerated without dose reduction for hematological toxicities. Olaparib must have been tolerated at a dose of 300mg twice daily for Arms A, B, & C. Olaparib must have been tolerated at a dose of 200 mg twice daily or higher for Arm D.

    For Cohort C and D Part II, patients may not have received cytotoxic chemotherapy in the interval between PARPi monotherapy and enrollment.
13. Patients who have had major surgery (as defined by the Site PI) must be fully recovered and ≥4 weeks post-operative prior to enrolling on study.
14. Patients must be able to swallow oral medications (capsules and tablets) without chewing, breaking, crushing, opening, or otherwise altering the product formulation. They should not have gastrointestinal illnesses that would preclude the absorption of AZD6738 or olaparib, which are oral agents.
15. Postmenopausal defined as:

    * Amenorrhea for 1 year or more following cessation of exogenous hormonal treatments;
    * LH and FSH levels in post-menopausal range for women under 50;
    * Radiation induced oophorectomy with last menses >1 year ago;
    * Chemotherapy-induced menopause with >1 yr interval since last menses;
    * Surgical sterilization (bilateral oophorectomy or hysterectomy).
16. Able to understand and voluntarily sign a written informed consent, and are willing and able to adhere to the protocol requirements.
17. Patients with a history of brain metastases diagnosed greater than one year prior to study entry may be considered if they received sterilizing therapy to the CNS (resection or radiation) and have been CNS recurrence-free for the one-year period.

Exclusion criteria:

1. Patients with known brain metastases diagnosed within one year will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
2. Patients who have had prior AZD6738 or other cell cycle checkpoint inhibitors such as other ATM or ATR inhibitor, WEE-1 inhibitor, or CHK1 (or 1/2) inhibitors.
3. Patients with a serious cardiac condition, such as congestive heart failure; New York Heart Association Class III/IV heart disease; unstable angina pectoris; myocardial infarction within the last 3 months; valvulopathy that is severe, moderate, or deemed clinically significant; or arrhythmias that are symptomatic or require treatment. Resting ECG with QTc > 470 msec on two or more time points within a 24-hour period or family history of long QT syndrome.
4. Patients with a systolic blood pressure <90 mm Hg at two consecutive visits or recurrent symptomatic orthostatic hypotension.
5. Lack of recovery of prior adverse events due to prior cancer therapy to Grade ≤1 (NCI CTCAE v5.0; except alopecia). Stable persistent Grade 2 peripheral neuropathy may be allowed as determined on a case-by-case basis at the discretion of the PI. Patients with platinum-related hypomagnesemia (on replacement) will be eligible.
6. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, clinically significant GI bleeding or hemoptysis within 28 days prior to the start of the study, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Another previous, active or current invasive malignancy within the last five years, with the exception of curatively treated stage IA cervical carcinoma, or resected stage IA, Grade 1 endometrial cancer, noninvasive non-melanoma skin cancers, DCIS of the breast or other solid tumors including lymphomas (without bone marrow involvement). Patients with localized breast cancer who are disease free at least three years out from treatment may be eligible.
8. Immunocompromised patients or HIV-positive patients on HAART due to potential drug interaction.
9. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is two weeks.
10. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is five weeks for enzalutamide or phenobarbital and three weeks for other agents.
11. Patients with myelodysplastic syndrome, acute myeloid leukemia, or with features suggestive of MDS/AML.
12. Major surgery within four weeks of starting study.
13. Patients with a known hypersensitivity to AZD6738 or olaparib or any of the excipients of the product.
14. Platinum refractory (progress in first line platinum therapy) are excluded for Cohorts A, B, C, D PART II.
15. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within three weeks prior to study treatment.
16. Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood and other body fluids.
17. Previous allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
18. Whole blood transfusions in the last 120 days prior to entry to the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecology Oncology trial for ovarian cancer patients.
Enrollment: 123 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 for all cohorts.
Response rate | 2 years
  Objective response rate (CR+PR) of the combination of AZD6738 and olaparib in women with recurrent ovarian cancer in platinum-sensitive and resistant, and PARP inhibitor resistant cohorts (e.g. Cohorts A, B, C, and D).

SECONDARY OUTCOMES:
Progression free survival | 2 years
  Clinical anti-tumor effect by standard criteria (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Simpkins, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided